CLINICAL TRIAL: NCT03884868
Title: Use of Iconographies for Risk Communication and Reduction of Patient's Anxiety During the Nurse Information Visit in the Colorectal Cancer Screening Program
Brief Title: Iconographies for Risk Communication and Reduction of Patient's Anxiety in a Colorectal Cancer Screening Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Pilar Lopez-Lopez, Principal Investigator, Corporacion Parc Tauli
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20198501
Record Dates: First submitted 2019-03-18; First posted 2019-03-21 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Colo-rectal Cancer
Keywords: Colorectal cancer screening; Iconographies; Risk communication; Patient medical knowledge
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Two consecutive study groups (no-concurrent).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Regular nursing visit: 1. Explanation of the meaning of a positive result in the FIT. 2. Explanation of the need to perform a colonoscopy with sedation. 3. Anamnesis. 4. Agreement of the day and hour to perform the colonoscopy. 5. Explanation of the diet and delivery of preparation for the preparation of the colon.
- Intervention group (Experimental): In addition of the regular nursing visit: the nurse will use iconographies specially designed to communicate the risk of the different possible diagnoses and the complications of the colonoscopy. Because the risks are different according to sex and age, specific iconographies will be developed from the data available in the first screening round.
  Interventions: Other: Iconographies to communicate risks

INTERVENTIONS:
Other: Iconographies to communicate risks — Use of iconographies to communicate the risks of the different possible diagnosis after a positive FIT during the screening program nurse visit.
  Arms: Intervention group

SUMMARY:
Background: Participants in the colon and rectal cancer (CRC) screening program that have a positive result in the Fecal Immunological Test (FIT) are visited by the screening nurse who explains the meaning of the positive test and the need to perform a colonoscopy. Having a positive result in the screening test can have a negative psychological impact on patients causing anguish.

Objective: To evaluate whether the use of iconographies to communicate the risks of possible diagnoses to patients with positive FIT improves the understanding of the information and reduces the degree of anguish.

Methods: Quasi-experimental pre-post intervention study with a control group. 240 individuals (men and women between 50-69 years of age, with a positive FIT result attending the nursing visit) will be included in two non-concurrent study groups (120 individuals per group). The control group will receive the nurse visit as usual. For the intervention group, the nurse will use iconographies to communicate the risk of the different possible diagnoses and the risk of complications of the colonoscopy. The degree of distress (Distress Thermometer and a scale of emotion-faces) will be measured before and after the visit and the understanding of the information (visual analog scale) after the visit. The degree of distress between the control group and intervention group will be compared.

If the results are favorable, the systematic use of iconographies can be implemented in the nursing screening visit and be extended to other Screening Units.

ELIGIBILITY:
Inclusion Criteria:

* women and men AND
* between 50 and 69 years of age AND
* who participate in the colorectal cancer screening program and have a positive result in the FIT AND
* who attend the nursing visit.

Exclusion Criteria:

* People who do not understand Catalan or Spanish OR
* with cognitive deterioration that prevents them from answering a questionnaire OR
* who do not know how to read or write.

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Grade of distress experienced by patients | Minute 0 (before the nurse visit)
  Grade of distress experienced by the patients measured with the Distress Thermometer (0-no distress to 10-high distress)
Grade of distress experienced by patients | at 30 minutes (after the nurse visit)
  Grade of distress experienced by the patients measured with the Distress Thermometer (0-no distress to 10-high distress)

SECONDARY OUTCOMES:
Grade of understanding of the information reported by patients | at 30 minutes (after the nurse visit)
  Grade of understanding of the information measured with a visual analogical scale (0-no understanding, 10- high understanding)

CONTACTS AND LOCATIONS:
Overall Officials: Pilar López-López, DUI, Principal Investigator — Corporació Sanitaria Parc Taulí
Locations (1):
- Parc Taulí Hospital Universitari, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No